CLINICAL TRIAL: NCT00820300
Title: An Open-Label, Phase 2 Study of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension (OH) or Open Angle Glaucoma (OAG)
Brief Title: A Safety Study of the Latanoprost Punctal Plug Delivery System (L-PPDS) in Subjects With Ocular Hypertension or Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 03
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Punctal plug (Experimental)
  Interventions: Drug: Latanoprost-PPDS

INTERVENTIONS:
Drug: Latanoprost-PPDS — Control of IOP compared to baseline for the experimental doses of Latanoprost-PPDS for 4 months or until loss of efficacy.

SUMMARY:
The purpose of this study is to determine if the Punctal Plug Delivery System is safe and effective in controlling intraocular pressure in patients with ocular hypertension or open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 yrs with ocular hypertension or open-angle glaucoma
* Subjects who have a best-corrected visual acuity of 20/100 or better.

Exclusion Criteria:

* Subjects who wear contact lenses.
* Uncontrolled medical conditions
* Subjects requiring chronic topical artificial tears, lubricants, and/or requiring any other chronic topical medications.
* Subjects who have a history of chronic or recurrent inflammatory eye disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzzani, MD, Study Director — QLT Inc.
Locations (1):
- Menlo Park, California, United States